CLINICAL TRIAL: NCT02619331
Title: Evaluation of High Speed Laser Doppler Imaging Technology to Quantify Skin Prick Tests in Allergic Volunteers
Brief Title: Evaluation of High Speed Laser Doppler Imaging Technology
Acronym: HSL-DI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, François Spertini, Associate Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSL-DI
Record Dates: First submitted 2015-07-30; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atopic volunteers (Experimental): Allergy tests will be performed in allergic patients with rhinoconjunctivitis and allergy test reading measured following two different methodologies. 1) test reading based on conventional wheal and flare measurement (wheal diameter in mm, CWFM), 2) test reading based on high speed laser doppler imaging (HS-LDI). Both type of tests reading will be compared.
  Interventions: Procedure: Allergy test reading

INTERVENTIONS:
Procedure: Allergy test reading — Reading of allergy skin tests (in response to allergen extracts or histamine or negative control) by HSL-DI versus direct observer evaluation (CWFM)

SUMMARY:
Skin prick tests (SPT) are commonly used in daily allergological practice to assess skin reactivity to allergens. Multiple factors can contribute to non-optimal results of conventional wheal and flare measurement (CWFM) of SPT such as inaccurate measurements, observer-dependency and absence of traceability.

This study aims to evaluate the quantification of SPT by a novel High Speed Laser Doppler Imaging (HSL-DI) and to compare it with CWFM. First, SPT with birch and/or grass pollen extracts as well as positive and negative controls will be performed in 20 volunteers (11 atopics, 9 non-atopics) to establish the characteristics (cut-off, optimal reading time and allergen concentration) of HSL-DI analysis based on two parameters ("area" and "flow" measurement). In a second step, fifty patients will be tested with birch and grass pollen extracts at optimal allergen concentration and time window. Analysis of SPT by HSL-DI and CWFM will be compared.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* history of allergic rhinitis to birch pollen and/or grass pollen.

Exclusion Criteria:

* any medical condition (including pregnancy) that could influence the study (viral or bacterial airway infection, active allergic rhinitis)
* uncontrolled asthma (peak expiratory "flow" <80% of volunteer's best personal value)
* treatment with antihistamine medication less than two weeks before enrolment or during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Skin microcirculation flow changes over time (composite autcome) | tests reading at 2.5 min., 5 min., 7.5 min., 10 min., 12.5 min., 15 min., 17.5 min. and 20 min.
  Skin microcirculation flow changes will be evaluated at 2.5 min., 5 min., 7.5 min., 10 min., 12.5 min., 15 min., 17.5 min. and 20 min. as measured in a composite outcome 1) by HS-LDI based on parameter "area" corresponding to the total number of non-zero pixels in the flare area and parameter "flow" as measured according to a specific formula in arbitrary units, or 2) as measured by conventional wheal and flare measurement (CWFM, direct observer reading) in mm.

CONTACTS AND LOCATIONS:
Overall Officials: François Spertini, MD, Principal Investigator — CHUV
Locations (1):
- CHUV , Division of Immunology and Allergy, Lausanne, Switzerland